CLINICAL TRIAL: NCT04699786
Title: Returning Research Results That Indicate Risk of Alzheimer Disease Dementia to Healthy Participants in Longitudinal Studies: Quantitative Analyses of a Randomized Clinical Trial
Brief Title: Returning Research Results That Indicate Risk of Alzheimer Disease Dementia to Healthy Participants in Longitudinal Studies
Acronym: WeSHARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202011119
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; Dementia of Alzheimer Type
Keywords: Dementia; Alzheimer disease dementia; genetics; neuroimaging
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Active Comparator): Participants randomized to Arm A will receive their research results two weeks after they review educational materials provided by the study and sign the informed consent document. Arm A is a neuroimaging arm.
  Interventions: Other: Arm A , Arm B, Arm C, & Arm D
- Arm B (Active Comparator): Participants randomized to Arm B will receive their research results one year after they review the educational materials provided by the study and sign the informed consent document. Arm B is a neuroimaging arm.
  Interventions: Other: Arm A , Arm B, Arm C, & Arm D
- Arm C (Active Comparator): Participants randomized to Arm C will receive their research results two weeks after they review educational materials provided by the study and sign the informed consent document. Arm C is a plasma amyloid arm.
  Interventions: Other: Arm A , Arm B, Arm C, & Arm D
- Arm D (Active Comparator): Participants randomized to Arm D will receive their research results one year after they review the educational materials provided by the study and sign the informed consent document. Arm D is a plasma amyloid arm.
  Interventions: Other: Arm A , Arm B, Arm C, & Arm D

INTERVENTIONS:
Other: Arm A , Arm B, Arm C, & Arm D — All arms will receive the same intervention, but at different time points. All arms will be offered the option to learn their research results in personalized five-year risk estimate of getting Alzheimer disease dementia. Arms A & C participants will receive their risk estimate about two weeks after consent is signed and Arms B& D will receive their risk estimate about one year after consent is signed. The risk estimate returned to participants is based on research results from individual genotyping results, imaging or plasma amyloid testing & demographic characteristics. All arms will complete psychosocial and cognitive testing. Also, surveys used in this study will ask about participants' experiences and feelings after learning their risk estimate. All arms will receive follow up calls at one week post disclosure of the risk estimate and surveys two, six, and twelve months post disclosure. Arms A & C will have extra surveys at twenty-four months post disclosure.

SUMMARY:
This is a study to evaluate the impact of returning research results that indicate a five-year risk estimate of Alzheimer disease dementia to participants without memory or thinking problems of the Knight Alzheimer Disease Research Center at Washington University in St. Louis.

DETAILED DESCRIPTION:
All participants without memory or thinking problems in a longitudinal observational cohort of aging (Memory and Aging Project) will be offered a five-year Alzheimer dementia risk estimate report that incorporates genetic and either neuroimaging research results or plasma amyloid results as well as demographic information into five-year Alzheimer disease dementia risk estimate. Using a two-year delayed-start randomized clinical trial design, participants will be randomized to receive research results either two weeks (Arm A/C) or one year (Arm B/D) after informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Current Knight ADRC participants who had their clinical assessment in the previous year.
* Minimum age of 65 years old
* Participant must be classified as cognitively normal (CDR® = 0) at their last clinical assessment.
* Participant has either recent research brain MRI and amyloid PET scan results, or recent plasma amyloid measurements (ideally within the past two years, but up to five years will be acceptable due to COVID-19-related delays).
* Participant has genetic research results available including APOE status.
* Participant is currently consented to be contacted for other research opportunities through the Knight ADRC.

Exclusion Criteria:

* There are no exclusion criteria, other than not meeting all of the inclusion criteria listed above.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Geriatric Depression Scale (GDS) | Based on parent study timeline. Measures are taken 12 months apart and straddle enrollment in trial. GDS is also measured at the time of informed consent.
  GDS is a questionnaire that screens for depression in older adults. It's a self-report tool that asks yes or no questions about how a person has been feeling over the past week.
Change in Clinical Dementia Rating sum of box score (CDR-SB) | Based on parent study timeline. Measures are taken 12 months apart and straddle enrollment in trial.
  Subjective measure of dementia determined as part of clinical assessment.
Change in cognitive composite score | Based on parent study timeline. Measures are taken 12 months apart and straddle enrollment in trial.
  Objective measure of cognitive functioning.

SECONDARY OUTCOMES:
Impact of Events Scale Revised (IES-R) | 2, 6, 12 and 24 months post-disclosure of risk estimate.
  A 15-item scale measuring distress specific to the test results received. Scores range from 0-75, with higher scores indicating greater test-related distress.
Decision Regret Scale | 2, 6, 12 and 24 months post-disclosure of risk estimate.
  The Decision Regret Scale measures "distress or remorse" after receiving research results.
Self- Report Heath Care Utilization | At consent, 6, 12 and 24 months post-disclosure of risk estimate
  This scale measures self-reported health care utilization that indicates both patients' health and their ability to self-manage their condition.
Understanding of Research Results | 2, 12 and 24 months post-disclosure of risk estimate.
  The scale measures participant's comprehension of their research results.
Patient Assessment of Communication Effectiveness | 2 months post-disclosure of risk estimate.
  This scale investigates participants' perspectives on communication and to measure how well the research team communicated research results to participants
Lifestyle/Health Behavior Change | 6, 12 and 24 months post-disclosure of risk estimate.
  This scale gauges self-reported preparedness of future health and end of life situations.
AD-Related Distress | At consent, 2, 6, 12 and 24 months post-disclosure of risk estimate.
  This scale measures participants' self-reported anxiety (psychological impact) about developing AD dementia.
Future Time Perspective | At consent, 12 and 24 months post-disclosure of risk estimate.
  This scale measures how participants' feel about future events and their self-reported agreement or disagreement with the future events.
Modified Social Impact Scale | 2, 6, 12 and 24 months post-disclosure of risk estimate.
  This scale assesses whether participant's self-image after learning research results indicating risk of developing AD dementia is affected by notions of stigma.
Views Regarding Research | At consent, 6 and 12 months post-disclosure of risk estimate.
  This scale assesses the impact of learning research results on attitudes towards research participation.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hartz, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data which documents, supports and validates research findings will be made available after the main findings from the final research data set have been accepted for publication. Such research data will be de-identified to prevent the disclosure of personal identifiers.
Supporting Information: SAP, Analytic Code
Time Frame: Data will be available immediately following publication with no end date.
Access Criteria: Access Criteria: Qualified researchers who provide a methodologically sound proposal will be able to access the data to achieve aims in the approved proposal.
  Proposals should be directed to hartzs@wustl.edu. To gain access, requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Hartz SM, Goswami S, Oliver A, Evans A, Jackson S, Linnenbringer E, Moulder KM, Morris JC, Mozersky J. What is the psychological and cognitive impact of returning Alzheimer disease dementia research results to healthy research participants? a delayed-start randomised clinical trial protocol for the WeSHARE study (Washington University study of having Alzheimer disease research results explained). BMJ Open. 2026 Jan 6;16(1):e099970. doi: 10.1136/bmjopen-2025-099970. PMID 41500647